CLINICAL TRIAL: NCT05500586
Title: The Effects of Glucagon on Hepatic Metabolism
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adrian Vella (Other)
Responsible Party: Sponsor-Investigator, Adrian Vella, Regulatory Sponsor, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22-000113
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Type2diabetes; NAFLD
Keywords: glucagon; insulin resistance; hepatic steatosis; amino acid metabolism
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Insulin Resistance; Fatty Liver | interventions — Glucagon

STUDY DESIGN:
Intervention Model Description: All subjects will undergo one study designed to measure the hepatic response to glucagon. There will be 3 groups non-diabetic and non-obese, obese, people with type 2 diabetes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy Adults (Experimental): We will study 20 subjects on one occasion using a hyperglycemic clamp with 2 doses of glucagon.
  Interventions: Drug: Glucagon response study
- Obese Adults (Experimental): We will study 20 subjects on one occasion using a hyperglycemic clamp with 2 doses of glucagon.
  Interventions: Drug: Glucagon response study
- Adults with Type 2 Diabetes (Experimental): We will study 20 subjects on one occasion using a hyperglycemic clamp with 2 doses of glucagon.
  Interventions: Drug: Glucagon response study

INTERVENTIONS:
Drug: Glucagon response study — Please see information in group descriptions
  Other Names: Glucagon

SUMMARY:
Whether impaired postprandial glucagon suppression in prediabetes and T2DM is an attempt to overcome resistance to glucagon's actions on hepatic AA catabolism, a defect in α-cell function, or a combination of both are important, unanswered questions. NAFLD is associated with T2DM risk and impaired insulin action. Unfortunately, it is unclear if glucagon resistance is caused by obesity, hepatic steatosis or both. The experiments outlined will determine if glucagon's actions on hepatic amino acid catabolism and EGP interact with hepatic lipid metabolism in lean and obese subjects with and without T2DM (and with varying degrees of hepatic steatosis).

DETAILED DESCRIPTION:
T2DM and prediabetes are characterized by abnormal post-prandial suppression of glucagon, which contributes to postprandial hyperglycemia by increasing EGP. Although these effects are magnified by decreased and delayed insulin secretion, they are also apparent when insulin secretion is intact. In rodents, altered glucagon signaling changes α-cell function and mass - an effect mediated by changes in circulating AA concentrations. Are the elevated concentrations of branched-chain AA and other AA metabolites in T2DM a cause or an effect of global α-cell dysfunction? Could altered glucagon signaling precipitate a vicious cycle resulting in T2DM?

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Able to give consent

Exclusion Criteria:

* History of prior upper abdominal surgery e.g. gastric banding, pyloroplasty, vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.
* Contraindications to MRI (e.g. metal implants, claustrophobia).
* Hematocrit < 35%
* TSH < 0.4 or > 5.5.
* Consumption of > 2 alcohol drinks per day or > 14 per week or a positive AUDIT questionnaire

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Amino acid catabolism in the presence / absence of glucagon | 240 minutes of study
  Tracer-dependent measurement of amino-acid clearance

SECONDARY OUTCOMES:
Effect of Diabetes on amino-acid catabolism | 240 minutes of study
  Tracer-dependent measurement of amino-acid clearance

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Derived] Christie HE, Mohan S, Egan AM, Boscolo F, Dalla Man C, Thompson SM, Jundt M, Fleming CJ, Andrews JC, Bailey KR, Jensen MD, Nair KS, Vella A. Hepatic steatosis in humans is associated with preserved glucagon action on amino acid metabolism. J Clin Invest. 2025 Dec 23:e200913. doi: 10.1172/JCI200913. Online ahead of print. PMID 41433112
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials